CLINICAL TRIAL: NCT01284231
Title: A Phase 1, Open-Label Study to Evaluate the Safety and Tolerability of MEDI-565 in Adults With Gastrointestinal Adenocarcinomas
Brief Title: A Study to Evaluate the Safety and Tolerability of MEDI-565 in Adults With Gastrointestinal Adenocarcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP216
Record Dates: First submitted 2011-01-18; First posted 2011-01-26 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Gastrointestinal Adenocarcinomas
Keywords: MEDI-565, gastrointestinal adenocarcinomas, carcinoembryonic antigen, bispecific T-cell engager

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MEDI-565 - Dose Escalation (Experimental): Up to 15 dose-escalation cohorts will be enrolled
  Interventions: Drug: MEDI-565
- MEDI-565 Dose Expansion Arm 1 (Experimental): 20 subjects with selected gastrointestinal tumor type will receive MEDI-565 at the maximum tolerated dose or optimum biologic dose
  Interventions: Drug: MEDI-565
- MEDI-565 Dose Expansion Arm 2 (Experimental): 20 subjects with selected gastrointestinal tumor type will receive MEDI-565 at the maximum tolerated dose or optimum biologic dose
  Interventions: Drug: MEDI-565
- MEDI-565 Dose Expansion Arm 3 (Experimental): Subjects with selected gastrointestinal tumor type will receive MEDI-565 at the maximum tolerated dose or optimum biological dose
  Interventions: Drug: MEDI-565

INTERVENTIONS:
Drug: MEDI-565 — MEDI-565 will be administered by IV infusion
  Arms: MEDI-565 - Dose Escalation
Drug: MEDI-565 — 20 subjects with selected gastrointestinal tumor type to receive MEDI-565 at the maximum tolerated dose or optimum biologic dose by IV infusion over 3 hours per day for 5 consecutive days every 28 days.
  Arms: MEDI-565 Dose Expansion Arm 1
Drug: MEDI-565 — 20 subjects with selected gastrointestinal tumor type to receive MEDI-565 at the maximum tolerated dose or optimum biologic dose by IV infusion over 3 hours per day for 5 consecutive days every 28 days.
  Arms: MEDI-565 Dose Expansion Arm 2
Drug: MEDI-565 — 20 Subjects with refractory Gastroesophageal cancer to receive MEDI-565 at the maximum tolerated dose or optimum biologic dose by IV infusion over 3 hours per day for 5 consecutive days every 28 days.
  Arms: MEDI-565 Dose Expansion Arm 3

SUMMARY:
To determine the maximum tolerated dose and/or optimum biologic dose of MEDI-565 in adult subjects and evaluate the safety profile in adult subjects with advanced gastrointestinal adenocarcinomas who have no available standard or curative treatments.

DETAILED DESCRIPTION:
This is a FTIH, dose-escalation and expansion Phase 1 study. The first part is a multicenter, open-label, single-arm, dose-escalation study of MEDI-565 to determine the MTD or OBD and evaluate the safety, tolerability, PK, IM, and antitumor activity of MEDI 565 in adult subjects who have GI adenocarcinomas for which no standard or curative treatments are available. The second part is a dose-expansion study at the MTD or OBD in subjects with selected tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age at the time of screening
* Adequate contraception from screening through end of trial
* For the dose-escalation phase, subjects with GI adenocarcinomas with no available standard or curative treatments
* Adequate hematological function
* Adequate organ function
* For subjects who had prior treatment with chemotherapy, biological therapy, radiotherapy, or had prior surgery: eligible for study entry if at least 30 days have passed since their treatment/surgery
* Life expectancy of at least 3 months
* Karnofsky performance status ≥ 70%
* Body weight ≥ 45 kg

Exclusion Criteria:

* Concurrent enrollment in another clinical study
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals
* Prior treatment with MEDI-565
* History of allergy or reaction to any component of the MEDI-565 formulation
* History of malignancy other than GI adenocarcinoma, within 5 years prior to study entry, with the exception of ductal carcinoma in situ of the breast, basal cell carcinoma of the skin or carcinoma in situ of the cervix successfully treated with curative therapy
* Diagnosis of hepatocellular carcinoma
* Clinical history of significant CNS pathology
* Active bacterial infection or known bacteremia.
* Vaccination within 2 weeks prior to initiation of MEDI-565
* Infection with HIV-1 or HIV-2; chronic infection with hepatitis B or C
* History of primary immunodeficiency
* History of chronic autoimmune disease
* Elective surgery planned during the study period through 30 days after discontinuation of MEDI-565.
* Treatment with any chemotherapy, radiotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment within 30 days prior to study entry and not recovered from treatment
* Treatment with any investigational agent within 30 days prior to initiation of MEDI-565
* Regular dose of systemic corticosteroids during the 30 days prior to initiation of MEDI-565 or anticipated need of corticosteroids exceeding prednisone 40 mg/day of prednisone or equivalent during the trial, or any other systemic immunosuppressive therapy within 30 days prior to study entry (some maintenance doses allowed)
* Contraindication to any protocol-specified concomitant medications administered during this study
* Pregnancy or lactation
* Evidence of any uncontrolled systemic disease (other than GI adenocarcinoma)
* Recent history of cardiac disease, including myocardial infarction, unstable angina pectoris or uncontrolled arrhythmia within 6 months, or evidence of severe congestive heart failure
* A marked baseline prolongation of corrected QT interval interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerable dose (MTD) or optimal biological dose (OBD) of MEDI-565 in subjects with gastrointestinal (GI) adenocarcinomas for which no standard or curative treatments are available. | MTD/OBD will be evaluated from the time of first administration of MEDI-565 through the first 28-day cycle
  MTD/OBD will be determined based on Dose Limiting Toxicities that will be evaluated from the time of first administration of MEDI-565 through the first 28-day cycle
Evaluate the safety profile in adult subjects with advanced gastrointestinal (GI) adenocarcinomas who have no available standard or curative treatments. | AEs and SAEs will be reported through 30 days after the last dose of MEDI 565
  The number (percentage) of subjects with AEs and SAEs reported through 30 days after the last dose of MEDI 565 will be summarized for all subjects who received at least one dose of study drug (Safety Population).

SECONDARY OUTCOMES:
Assess the safety and antitumor activity of MEDI-565 in the dose-expansion phase. | 3 years
  The antitumor activity of MED-565 will be assessed using objective response rate (ORR), time to response (TTR), duration of response (DR), time to progression (TTP), progression-free survival (PFS), and overall survival (OS) using RECIST guidelines
Pharmacokinetics of MEDI-565 | 3 years
  Individual MEDI-565 concentrations will be tabulated by dose cohort along with descriptive statistics. Noncompartmental PK data analysis will be performed for data obtained from each dose cohort with scheduled PK sample collection. If the data allow, descriptive statistics of noncompartmental PK parameters (AUC, Cmax, Tmax, CL, Vd, t½) will be provided.
Immunogenicity of MED-565 | 3 years
  The immunogenic potential of MEDI-565 will be assessed by summarizing the number and percentage of subjects who develop detectable anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McDevitt, Study Director — MedImmune LLC
Locations (4):
- United States (4):
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Augusta, Georgia
  - Research Site, Durham, North Carolina
  - Research Site, Philadelphia, Pennsylvania